CLINICAL TRIAL: NCT00001430
Title: A Randomized Study of EPOCH II Versus EPOCH II and Immunotherapy in Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 950073; 95-C-0073
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-01

CONDITIONS: Hodgkin's Disease; Non Hodgkin's Lymphoma
Keywords: IL-2; Drug Resistance; Continuous Infusion; Peripheral Stem Cells; MDR
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Interleukin-2

INTERVENTIONS:
Procedure: PBSC
Drug: IL-2
Drug: EPOCH II

SUMMARY:
This is a randomized study of combination chemotherapy (EPOCH II) versus EPOCH II and immunotherapy with peripheral blood stem cells (PBSC) and IL-2 in patients with relapsed Hodgkin's and non-Hodgkin's lymphomas, and untreated patients with low-grade non-Hodgkin's lymphomas. The chemotherapy entails the administration of multiple cycles of infusional doxorubicin, etoposide and vincristine chemotherapy (total of 3), alternating with cycles of high-dose cyclophosphamide (3 cycles). Patients will be randomized, on a 2:1 basis, to either receive only chemotherapy or to undergo a PBSC harvest with PBSC reinfusion and IL-2 following the last cycle of chemotherapy. In all patients, immunological monitoring for NK/LAK activity, T cell number and function will be performed. The therapy is specifically targeted for patients who would be candidates for high-dose chemotherapy with stem cell support.

DETAILED DESCRIPTION:
This is a randomized study of combination chemotherapy (EPOCH II) versus EPOCH II and immunotherapy with peripheral blood stem cells (PBSC) and IL-2 in patients with relapsed Hodgkin's and non-Hodgkin's lymphomas, and untreated patients with low-grade non-Hodgkin's lymphomas. The chemotherapy entails the administration of multiple cycles of infusional doxorubicin, etoposide and vincristine chemotherapy (total of 3), alternating with cycles of high-dose cyclophosphamide (3 cycles). Patients will be randomized, on a 2:1 basis, to either receive only chemotherapy or to undergo a PBSC harvest with PBSC reinfusion and IL-2 following the last cycle of chemotherapy. In all patients, immunological monitoring for NK/LAK activity, T cell number and function will be performed. The therapy is specifically targeted for patients who would be candidates for high-dose chemotherapy with stem cell support.

ELIGIBILITY:
Patients must be between 18 and 70 years old.

All stages of patients with low-, intermediate- or high-grade non-Hodgkin's lymphomas, or Hodgkin's disease who have disease following standard chemotherapy.

Stage II-IV patients with previously untreated low-grade lymphoma or untreated low-grade with progression.

Patients must have received less than or equal to 2 prior combination chemotherapy regimens, no combination chemotherapy refractory disease, no high-dose chemotherapy with stem cell rescue, and may not have CNS involvement by lymphoma.

Pathology slides must be reviewed and a diagnosis of lymphoma confirmed by the Hematopathology Section, Laboratory of Pathology, NCI.

No patients with a history of coronary artery disease with angina pectoris and/or an ejection fraction less than 42 percent.

Serum creatinine clearance greater than 50 cc/min, bilirubin less than 2.5 u and AST/ALT less than 2x normal, absolute neutrophil count greater than 1000/mm(3) and platelet count greater than or equal to 100,000/mm(3) unless due to respective organ involvement by tumor.

Patients must have an ECOG performance status less than or equal to 2.

Patients must be HIV negative.

Pregnant women will be excluded.

Patients must be able to give informed consent.

Patients who, in the opinion of the principal investigator, are poor psychiatric or medical risks because of non-malignant systemic disease will be excluded.

A completed eligibility form.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49
Dates: Start 1995-02; Study Completion 2002-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Wilson WH, Bryant G, Bates S, Fojo A, Wittes RE, Steinberg SM, Kohler DR, Jaffe ES, Herdt J, Cheson BD, et al. EPOCH chemotherapy: toxicity and efficacy in relapsed and refractory non-Hodgkin's lymphoma. J Clin Oncol. 1993 Aug;11(8):1573-82. doi: 10.1200/JCO.1993.11.8.1573. PMID 7687667
- [Background] Vose JM, Anderson JR, Kessinger A, Bierman PJ, Coccia P, Reed EC, Gordon B, Armitage JO. High-dose chemotherapy and autologous hematopoietic stem-cell transplantation for aggressive non-Hodgkin's lymphoma. J Clin Oncol. 1993 Oct;11(10):1846-51. doi: 10.1200/JCO.1993.11.10.1846. PMID 8105034
- [Background] Mackall CL, Granger L, Sheard MA, Cepeda R, Gress RE. T-cell regeneration after bone marrow transplantation: differential CD45 isoform expression on thymic-derived versus thymic-independent progeny. Blood. 1993 Oct 15;82(8):2585-94. PMID 7691265